CLINICAL TRIAL: NCT02637271
Title: Neural Correlates of a Nutritionally Balanced Total Meal Replacement, 3 Week Dietary Exposure: An fMRI Study
Brief Title: Brain Response to Dietary Interventions
Acronym: BRDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 109416/A16-0067-001
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: Calorie restriction; Meal replacement; fMRI; Food-cue reactivity; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Meal Replacement (Experimental): Participants will be provided instruction in the appropriate use of the meal replacement product. The participants will be directed to refrain from all items of food for a period of 21 days except for the meal replacement products and vitamin supplements provided by the investigators (1120 kcal/day). Optifast™ 800 total meal replacement shakes will be provided to the participants for the 21 day intervention period.
  Interventions: Other: Low calorie total meal replacement
- Typical Diet (Active Comparator): Participants will be directed to use portion control to maintain a calorie level no greater than 1120 kcal per day. The participants will be directed to continue to consume food and beverage items that are representative of their typical diet (with the exception of reduced portions). Participants will be provided resources to assist them in determining caloric content of foods eaten.
  Interventions: Other: Low calorie typical diet

INTERVENTIONS:
Other: Low calorie total meal replacement — Participants will be provided instruction in the appropriate use of the meal replacement product. The participants will be directed to refrain from all items of food for a period of 21 days except for the meal replacement products and vitamin supplements provided by the investigators (1120 kcal/day). Optifast™ 800 total meal replacement shakes will be provided to the participants for the 21 day intervention period.
  Arms: Total Meal Replacement
Other: Low calorie typical diet — Participants will be directed to use portion control to maintain a calorie level no greater than 1120 kcal per day. The participants will be directed to continue to consume food and beverage items that are representative of their typical diet (with the exception of reduced portions). Participants will be provided resources to assist them in determining caloric content of foods eaten.
  Arms: Typical Diet

SUMMARY:
In order to better understand how commonly used dietary interventions for obesity influence brain activity and in turn people's ability to adhere to their healthy nutrition plan, the investigators need to study how people's brains react to food cues while undergoing such interventions. Our study will add to our understanding of neural (brain) regulation of hedonic and homeostatic mechanisms (i.e. pleasure and hunger) in influencing adherence to calorie-reduced eating plans.

DETAILED DESCRIPTION:
Recruitment of subjects: Advertisements for the recruitment of participants will be posted on social media and notice boards within the Texas Tech University (TTU) including the web-based notice boards (including but not limited to Tech Announce, Craig's List). Announcements will also be made using the same materials targeting the local community through paid advertisement in local print and online media outlets (e.g. newspapers) and through flyers distributed within area medical clinics and fitness centers. Thirty-two obese (BMI > 30) male and female subjects will be enrolled with the intended completion of at least 30 (15 per group).

Pre-Screening (Telephone): Individuals who express an interest in participating will be contacted by a graduate or undergraduate research assistant who will administer a structured telephone interview to: 1) provide information related to the requirements of the study, along with potential risks and benefits 2) Screen for eligibility based on specific inclusion and exclusion criteria. All potential subjects will be informed that their responses will remain confidential and that taking part in the screening interview in no way obligates them to participate.

Potential participants who meet participation criteria as assessed via the telephone prescreening process will be contacted by the study team via email/phone within 48 hours following the interview to inform of eligibility (or ineligibility) and to schedule an initial, in person assessment (Visit 1) if deemed eligible.

Visit 1 (Screening and Consent): This in-person screening visit will include the following: Participants will be provided with the Behavioral Medicine and Translational Research (BMTR) Health & Weight History Form to complete upon arrival at the clinic. Weight, height, BMI and body fat percentage via bio-electrical impedance analysis (BIA) using the TANITA BC-418 segmental body composition analyzer (TANITA Corporation of America Inc., IL, USA) and body composition analysis unit; measured blood pressure (BP) via Omron Digital BP Monitor HEM-907XL (Omron Healthcare Inc., IL, USA) will be obtained.

If inclusion/exclusion criteria are met; informed consent will be obtained and the participant will be considered 'enrolled' in the study at that time. Participants will be scheduled for 2 scanning visits (visits 2 and 5) and the 2 check in visits (visits 3 and 4) at this time and instructed on the procedures for these subsequent visits. At completion of Visit 1 the participants will be told to make no deviation from their standard diet until after their initial fMRI scan visit (visit 2).

Special Scheduling Considerations: The phase of the menstrual cycle may have an effect on cravings. The first scanning session of pre-menopausal female participants will be scheduled in the second half of the follicular phase of a menstrual cycle (i.e. 10th - 14th day of a menstrual cycle). Thus, the second scanning session, which will be performed 3 weeks after the first session, will be performed in the first half of the follicular phase (approximately between the 3rd and 7th days) of the next menstrual cycle. This will ensure that both scanning sessions will be performed within the follicular phase.

Visit 2 (Pre-intervention fMRI Scan):

1. Participants will be requested to refrain from taking any items of food or beverages (except water) for 8 hours minimum prior to the scanner visit.
2. The participants will also be advised to refrain from i) tobacco use in any form ii) the intake of alcohol or caffeine in any form within the 24 hours prior to the scanning visit.
3. The participants will be asked to complete the following paper & pencil measures in an adjacent room prior to entering the fMRI scanner: i) Food Craving Inventory; ii) Power of Food Scale; iii) Three-Factor Eating Questionnaire; iv) Yale Food Addiction Scale; v) Visual Analogue Scales (VAS) on the dimensions of hunger, satiety, thirst, fullness and emptiness.
4. The duration of each scan will be 45-60 minutes (including the time spent on placing each participant in the scanner).
5. After the scanning is complete, each participant will be taken to an adjacent room and VAS will be administered again immediately after the scan (total duration 30 minutes) according to the procedures outlined in (c) above.
6. The participants will then be shown on a laptop computer, a random subset of 60 images from the set to which the participants were exposed to, during the fMRI scanning paradigm, randomly mixed with 60 other images to which the participants were not exposed with a task of recognizing the images that were presented in the scanning paradigm (duration 15-20 minutes).

fMRI scanning paradigm: An event-related design will be used for all stimulus presentations. 120 images of two categories (food items and objects) will be displayed on an LCD screen and projected via a mirror attached to the head coil. Images of food and objects will be matched for contrast, brightness, size and resolution. Food images will represent a continuous spectrum of highly rewarding to less rewarding items, while selected common objects (e.g. a paper clip) will be deemed 'neutral'. Each participant will be shown a fixation cross lasting for 2000-4000ms. Then, each visual image will be presented for 5000-6000ms with 'overlapped' opportunity for rating of the stimulus by the subject (i.e., ratings performed while viewing the image). During the presentation of each image, participants will be required to answer the question "How much do you want it now?" on a 1-7 Likert scale using fiber optic buttons. This sequence will be conducted 30 times, with different images to complete each run. Eight such runs will comprise each scanning session. Following the stimulus presentation phase (EPI scan), a T1-weighted structural scan (SS) lasting approximately 5 minutes will be obtained followed by a diffusion tensor imaging (DTI) scan (6 minutes) to assess white-matter connectivity.

Immediately following the initial fMRI scan subjects will be randomly assigned to one of the 2 arms of the study: the Total Meal Replacement (TMR) group or the Typical Diet (TD) group (16 participants per group). Each arm will maintain 1120 kcal/day target caloric intake.

TMR Group: Optifast™ 800 total meal replacement shakes (1120 kcal/day) will provide all nutrition (no additional food). One week supply of meal replacement product is provided.

TD Group: Participants will be directed to use portion control to maintain a calorie level of 1120 kcal per day. Subjects will be provided resources to assist them in determining caloric content of foods eaten.

Visits 3 and 4 (Check-in Visits): Subjects of both groups will be requested to return to the BMTR lab at 1 week intervals over the first 2 weeks following visit 2 to be weighed, have blood pressure taken, review any issues and report adherence variations from protocol (including additional caloric intake). Subjects of the TMR group will receive the next week's product at each visit. Subjects of the TD group will be requested to provide a written list of daily calorie intake of the past week at each visit.

Visit 5 (post-intervention Scanning Visit): Preparation for the visit, completion of pencil and paper measures, procedure of scanning and the post-scan memory task will be similar to visit 2. In addition, BIA, BP, weight and height will be measured and BMI will be calculated.

Analysis: fMRI analysis will be carried out using a standard mixed effects model implemented in FMRIB Software Library (FSL). Specifically, analysis of fMRI data will be focused on identifying pre-post differences in both the location and relative magnitude of whole brain activation patterns within and between members of each group (TMR vs. TD). Pre-planned comparisons will also be made for specific regions of interest: a) food-reward related areas (e.g. insula, orbito-frontal cortex, anterior cingulate cortex, and amygdala); b) reward calculating regions (e.g. nucleus accumbens and ventral striatum), c) memory and emotion related areas (e.g. hippocampus and amygdala); d) homeostatic circuitry (i.e. hypothalamus) and cortical areas exerting executive control (e.g. pre-frontal cortex). Both structural and functional connectivity between the considered regions of interest will also be modeled and compared between and within groups. Demographic, health, weight history and psychosocial variables may be included as covariates in specific analyses as indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19-60 years
2. BMI of 30-39.9 kg/m2 (upper limit due to scanner comfort/feasibility)

Exclusion Criteria:

1. Participants unable to provide informed consent.
2. Participants with motor, visual or hearing impairment.
3. Females with irregular menstrual cycles.
4. Patients currently diagnosed with diabetes mellitus, experiencing uncontrolled hypertension, history of ischemic heart disease, cerebrovascular accidents, neurological disease or current severe psychiatric illness (e.g. psychosis, schizophrenia, severe untreated depression, current suicidal ideation, and current or past suicide attempts), history of psychiatric hospitalization.
5. Women who are pregnant or who are attempting to conceive.
6. Participants with contraindications for fMRI scanning.

   * aneurism clips
   * any implanted medical devices (pacemaker, neurostimulator)
   * known pregnancy
   * shrapnel in body or any injury to eye involving metal
   * any ferrous metal in body
7. Participants with a history of eating disorders such as bulimia nervosa, anorexia nervosa and severe binge eating disorder.
8. Participants with a history of substance abuse or alcohol abuse.
9. Participants who are currently on or have been on within the past 4 weeks any anti-depressant, anti-epileptic, or anxiolytic medicines.
10. Patients experiencing persistent loss of appetite, nausea or vomiting within the last 4 weeks.
11. Participants who have been involved in a weight loss intervention program (including anti-obesity medication) within the past 3 months or who have had bariatric surgery.
12. Current smokers (within the last 30 days).

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in fMRI Food-cue Reactivity | Baseline (pre-intervention) and 3 weeks (post-intervention)

SECONDARY OUTCOMES:
Change in sub-scales of the Food Craving Inventory | Baseline (pre-intervention) and 3 weeks (post-intervention)
Change in sub-scales of the Three-factor Eating Questionnaire | Baseline (pre-intervention) and 3 weeks (post-intervention)
Change in Power of Food Scale | Baseline (pre-intervention) and 3 weeks (post-intervention)
Change in Yale Food Addiction Scale | Baseline (pre-intervention) and 3 weeks (post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, PhD, Principal Investigator — Texas Tech University - Department of Nutritional Sciences
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dye L, Warner P, Bancroft J. Food craving during the menstrual cycle and its relationship to stress, happiness of relationship and depression; a preliminary enquiry. J Affect Disord. 1995 Jun 8;34(3):157-64. doi: 10.1016/0165-0327(95)00013-d. PMID 7560543
- [Background] White MA, Whisenhunt BL, Williamson DA, Greenway FL, Netemeyer RG. Development and validation of the food-craving inventory. Obes Res. 2002 Feb;10(2):107-14. doi: 10.1038/oby.2002.17. PMID 11836456
- [Background] Lowe MR, Butryn ML, Didie ER, Annunziato RA, Thomas JG, Crerand CE, Ochner CN, Coletta MC, Bellace D, Wallaert M, Halford J. The Power of Food Scale. A new measure of the psychological influence of the food environment. Appetite. 2009 Aug;53(1):114-8. doi: 10.1016/j.appet.2009.05.016. Epub 2009 Jun 12. PMID 19500623
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale. Appetite. 2009 Apr;52(2):430-6. doi: 10.1016/j.appet.2008.12.003. Epub 2008 Dec 11. PMID 19121351
- [Derived] Kahathuduwa CN, Davis T, O'Boyle M, Binks M. Do scores on the Food Craving Inventory and Three-Factor Eating Questionnaire correlate with expected brain regions of interest in people with obesity? Physiol Behav. 2018 May 1;188:1-10. doi: 10.1016/j.physbeh.2018.01.018. Epub 2018 Feb 3. PMID 29421336